CLINICAL TRIAL: NCT07124637
Title: Investigating the Effect of an Educational Intervention Based on Social Cognitive Theory on Promoting Fruit and Vegetable Consumption Among Students
Brief Title: Educational Intervention on Promoting Fruit and Vegetable Consumption Among Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arash Salahshouri, Faculty member, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IR.AJUMS.REC.1402.106
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Promoting on Fruit and Vegetable Consumption
Keywords: Fruit; Vegetables; healthy nutrition; educational intervention; Social Cognitive Theory

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group design, where participants are assigned to one of two groups: an intervention group or a control group. Each group was followed concurrently throughout the study period. The intervention group receives a multilevel blended educational program based on Social Cognitive Theory, while the control group does not receive this program. Outcomes related to fruit and vegetable consumption and cognitive-social constructs were measured and compared between groups at baseline and two months after the intervention. This design allows for direct comparison of the intervention's effectiveness against usual conditions without intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention Group (Experimental): Female students in grades 7-9 received a multilevel educational intervention based on Social Cognitive Theory to increase fruit and vegetable consumption. The program included seven 60-minute sessions that were delivered both face-to-face at schools and virtually via WhatsApp, focusing on enhancing constructs of Social Cognitive Theory. Parents received online training and supportive text messages. School staff cooperated to improve access to fruits and vegetables and displayed educational materials to reinforce behavior change.
  Interventions: Behavioral: Multicomponent Social Cognitive Theory-Based Educational Program to Increase Fruit and Vegetable consumption in Students
- Arm 2: Control Group (No Intervention): Participants in this arm are female students in grades 7 to 9 who do not receive any educational intervention during the study period. They complete the same baseline and follow-up assessments as the intervention group but continue their usual activities without additional programs related to diet or nutrition.
  Intervention Details:
  No intervention provided Participate in data collection before and two months after the intervention period.

INTERVENTIONS:
Behavioral: Multicomponent Social Cognitive Theory-Based Educational Program to Increase Fruit and Vegetable consumption in Students — This multilevel blended educational intervention applies Social Cognitive Theory (SCT) to increase fruit/vegetable (F/V) intake among female middle school students. The 8-week program includes:
  A) Student Components:
  * Seven 60-minute sessions (4 in-person, 3 WhatsApp-delivered)
  * Interactive activities: cooking demonstrations, goal-setting workshops, and educational games
  * SCT-focused content: self-efficacy building, outcome expectation modification
  B) Parental Engagement:
  * Weekly SMS nutrition tips
  * Two virtual workshops on creating F/V-supportive home environments
  * School Environment Modifications:
  * Cafeteria redesign to promote F/V accessibility
  * Peer-led 'Healthy Eating Ambassador' program
  Unique aspects distinguishing this intervention:
  * First SCT-based program specifically adapted for Iranian adolescent females
  * Dual delivery (in-person + digital) optimized for school settings
  * Simultaneously targets individual, social, and environmental determinants.
  Arms: Arm 1: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if a multilevel blended educational intervention based on Social Cognitive Theory (SCT) can increase fruit and vegetable (F&V) consumption among female students.

The main questions it aims to answer are:

* Does an SCT-based educational program increase the daily amount of fruit and vegetable intake among adolescent girls?
* Does the intervention improve key cognitive-social constructs such as self-efficacy, self-regulation, knowledge, behavioral skills, and social support related to healthy eating? Researchers will compare students in the intervention group who receive seven 60-minute blended sessions (including face-to-face and WhatsApp-based education) tailored according to SCT constructs to a control group receiving no intervention.

Participants will:

* Attend scheduled educational sessions covering nutrition knowledge, skill-building (e.g., meal preparation with F&V), and behavior change strategies.
* Participate in activities designed to enhance self-efficacy, observational learning, and social support for healthy eating.
* Complete validated questionnaires assessing F&V intake and SCT-related cognitive-social constructs before and two months after the intervention.

This study evaluates whether integrating theory-driven, multilevel interventions in schools is effective in promoting healthier dietary habits among adolescent girls, especially in a resource-constrained setting.

DETAILED DESCRIPTION:
This cluster-randomized controlled trial was conducted from April 2023 to October 2024 in four public middle schools in Seydun, Khuzestan Province, Iran. The primary aim was to evaluate the effectiveness of a multilevel blended educational intervention based on Social Cognitive Theory (SCT) in increasing fruit and vegetable (F&V) consumption among female students in grades 7 to 9.

Study Design and Setting:

A two-group parallel design was employed. Four public middle schools in Seydun were randomly assigned by cluster randomization: two schools to the intervention arm and two schools to the control arm. This design minimized contamination and strengthened internal validity. The intervention spanned eight weeks, delivered through a blended format combining in-person sessions and virtual meetings via WhatsApp.

Participants and Sampling:

The target population included all female students in grades 7, 8, and 9 attending the selected schools. Multistage sampling was performed. Initially, schools were randomly chosen, and then from each grade, students were selected by convenience sampling to reach the calculated sample size. Eligibility criteria included absence of nutrition-related diseases (such as diabetes or morbid obesity), no participation in concurrent similar educational programs, smartphone access for virtual components, residency in Seydun city, and provision of informed consent by both students and their parents.

A total of 252 students were initially enrolled (126 in each arm). Following attrition due to withdrawal, incomplete questionnaires, and other reasons, 205 participants completed the study (104 in intervention, 101 in control).

Intervention:

The intervention was designed and implemented based on the Social Cognitive Theory framework, targeting multiple levels of influence on dietary behaviors including individual cognition, social support, and environmental conditions.

Seven 60-minute sessions were delivered over approximately two months. These sessions employed various teaching methods: lectures, group discussions, Q&A, drawing activities, audiovisual clips, small texts, slides, posters, and pamphlets. Content was tailored using baseline pre-test data and SCT constructs such as self-efficacy, self-regulation, outcome expectations and values, behavioral skills, observational learning, environmental influences, and social support.

In addition to direct education, the program worked collaboratively with parents and school staff. Parent workshops emphasized creating a supportive home environment by encouraging regular provision of fresh fruits and vegetables and reducing availability of unhealthy snacks. School cafeteria staff were engaged to improve accessibility to healthy food options. Student groups promoting healthy eating were also formed to foster peer support and positive norms.

The control group received no educational intervention but completed baseline and follow-up questionnaires at similar time intervals.

Data Collection Instruments:

Data were collected using a comprehensive, researcher-developed questionnaire validated for this population. It comprised:

Demographic and background characteristics (age, BMI, parental education and occupation, household income, etc.) Dietary intake frequency of various fruits and vegetables measured on a 6-point scale (0 = none to 5 = 5 or more servings per day)

* SCT constructs assessed by multiple scales:
* Self-efficacy (6 items)
* Self-regulation (4 items)
* Observational learning (4 items)
* Outcome expectations (9 items)
* Outcome values (7 items)
* Knowledge (14 items with multiple-choice and true/false questions)
* Behavioral skills (3 items)
* Environmental conditions (8 items)
* Social support (4 items) Responses used Likert scales ranging from 1 (strongly disagree/never) to 5 (strongly agree/always). The questionnaire demonstrated high validity and reliability (Cronbach's alpha = 0.92).

Procedures:

After obtaining ethics committee approval, informed consent was secured. Baseline data collection was conducted before the intervention in both groups. The intervention group participated in the blended educational program while the control group did not receive education.

Follow-up data collection occurred two months post-intervention using the same questionnaire tools. Data quality control included filtering incomplete questionnaires, answer time thresholds to ensure validity, and attrition monitoring.

Statistical Analysis:

Data normality was tested using Kolmogorov-Smirnov tests. Descriptive statistics summarized participant characteristics. Chi-square and Fisher's exact tests compared categorical variables between groups. Independent t-tests assessed intergroup differences in quantitative measures. Paired t-tests evaluated within-group changes. Analysis of covariance (ANCOVA) was performed to adjust for baseline differences when assessing intervention effects on F&V consumption.

ELIGIBILITY:
Inclusion Criteria:

* Free of nutrition-related diseases,
* Not following any special diets or weight loss programs,
* Provided informed consent to participate,
* Possess a smartphone compatible with the educational application,
* Residents of Seydun city,
* Not currently participating in similar educational programs.

Exclusion Criteria:

* Incomplete or invalid questionnaire responses (e.g., response time less than 7 minutes),
* Absence from more than one educational session,
* Voluntary withdrawal from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-05-12 (Actual)

PRIMARY OUTCOMES:
Change in Daily Fruit and Vegetable (F&V) Consumption | Baseline (pre-intervention) and 2 months post-intervention.
  Daily fruit and vegetable consumption among female students in grades 7 to 9 was assessed using a validated dietary questionnaire. This researcher-developed instrument included 27 items across two sections-12 items for fruit and 15 items for vegetable intake-measured on a 6-point scale ranging from 0 ("Did not consume") to 5 ("5 servings per day"). Consumption was expressed as the average number of daily servings, with scores ranging from 0 to 5. Higher scores indicate greater F&V intake, reflecting healthier dietary behavior.

SECONDARY OUTCOMES:
Changes in Cognitive-Social Determinants Related to Fruit and Vegetable Consumption | Before and two months after the intervention.
  This outcome assesses changes in Social Cognitive Theory (SCT)-based determinants of fruit and vegetable intake, including self-efficacy (6 items; Self-Efficacy Scale for fruit and vegetable consumption, score range: 6-30), self-regulation (4 items; score range: 4-20), observational learning (4 items; score range: 4-20), outcome expectations (9 items; score range: 9-45), outcome values (7 items; score range: 7-35), knowledge (14 items; score range: 0-14), and behavioral skills (3 items; score range: 3-15). On all scales, higher scores indicate more favorable outcomes, such as greater self-efficacy or higher knowledge levels. These constructs were measured using validated questionnaires at baseline and two months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Salahshouri, Ph.D., Principal Investigator — Ahvaz Jundishapur University of Medical Sciences
Locations (1):
- Seydun Public Schools, Ahvāz, Khouzestan, Iran

IPD SHARING:
Plan to Share IPD: Undecided
Public release of these data is not part of the research plan. However, upon reasonable request from researchers, and with ethics committee approval and strict confidentiality maintained, participant data can be shared with researchers in a controlled and limited manner.